CLINICAL TRIAL: NCT01251770
Title: Variation in Natremia Using Two Different Maintenance Intravenous Fluids in Postsurgical Hospitalized Children
Acronym: surgical-Na
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HGNPE-15-2010
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2012-01-25 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Hyponatremia
Keywords: Hyponatremia; Water-Electrolyte Imbalance
MeSH Terms: conditions — Hyponatremia; Water-Electrolyte Imbalance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- half saline (Experimental): Subjects in this arm will receive 0.45% NaCl/dextrose 5% intravenous (IV) maintenance fluids.
  Interventions: Drug: 0.45% NaCl/dextrose 5%
- third saline (Active Comparator): Subjects in this arm will receive 0.3% NaCl/dextrose 5% intravenous (IV) maintenance fluids.
  Interventions: Drug: 0.3% NaCl/dextrose 5%

INTERVENTIONS:
Drug: 0.45% NaCl/dextrose 5% — Subjects in this arm will receive 0.45% NaCl/dextrose 5% intravenous (IV) maintenance fluids.Total daily fluid infusion equal to: 80 ml/kg/day for those weighing up to 10 kg, and 1500 ml/m^2 body surface.
  Other Names: half saline
  Arms: half saline
Drug: 0.3% NaCl/dextrose 5% — Drug: 0.3% NaCl/dextrose 5% IV maintenance fluids. Total daily fluid infusion equal to: 80 ml/kg/day for those weighing up to 10 kg, and 1500 ml/m^2 surface.
  Other Names: third saline
  Arms: third saline

SUMMARY:
The primary objective of this study is to compare the blood sodium level after 12 hours following the initiation of therapy with either 0.3% NaCl/dextrose 5% or 0.45% NaCl/dextrose 5%, in postsurgical hospitalized children requiring maintenance IV fluid administration.

DETAILED DESCRIPTION:
Background: Despite prescription of maintenance IV fluids in hospitalized children is widely used since 1957 (Holiday & Segar), it is not always adequate for children with acute diseases, leading to hyponatremia. This mainly occurs due to a non-physiologic ADH secretion in this group of patients due to nausea, stress, pain, and surgical interventions, and the use of hypotonic maintenance IV fluids.

0.3% NaCl/dextrose 5%, is widely use as IV maintenance fluid in children after surgery. There is evidence suggesting that these IV fluids used in postsurgical hospitalized patients do not provide the adequate amount of sodium they require, leading to an increased risk of developing hyponatremia. Using 0.45% NaCl/dextrose 5% as IV maintenance fluid in these children would prevent hyponatremia, but this treatment has not been totally studied yet.

Study procedures: Hospitalized children who fulfill inclusion criteria and not having any of the exclusion criteria will be considered for the enrolment after written informed consent.

Venous blood samples will be taken at enrollment (baseline) for estimation of serum sodium. After randomization, one group will receive 0.3% NaCl/dextrose 5%, IV, at standard maintenance rate (100 ml/kg for the first 10 kg of body weight, 50 ml/kg for the next 10 kg, and 20 ml/kg for body weight exceeding 20 kg). The second group will receive 0.45% NaCl/dextrose 5%, IV, at the same rate.

Serum sodium will be estimated in both groups after 12 hours of intravenous fluid therapy.

Children who required oral fluids will be excluded from per-protocol analysis, and only analyzed for intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Postsurgical children admitted to HGNPE Department of Surgery between january 2010 and october 2011.

Aged 1 month to 16 years. Initial plasma Na between 135-145 mmol/L. Primary route of fluid administration is anticipated to be intravenous, in the first 12 hours following surgery.

Informed consent of parent/guardian.

Exclusion Criteria:

* • Children with illness that have primary fluid and electrolyte imbalance such as:

  * Shock: Defined as acute circulatory failure resulting in decreased tissue perfusion and manifesting as altered sensorium, hypothermia (<35oC), tachycardia, prolonged capillary filling time (>3 seconds), hypotension (BP < 5th percentile for age), oliguria (<0.5 ml/kg/hr), hypoxemia, hyperlactatemia, requirement of fluid bolus and/ or vasopressors.
  * Diarrhea and Dehydration: Children presenting with diarrhea and features of dehydration: lethargy, irritability and altered sensorium, thirst, decreased urine output, sunken eyes & dry mucous membranes, loss of skin elasticity.; children with ongoing diarrhea will be excluded even if there is no dehydration.
  * Fluid Overload: Cirrhosis, Congestive heart failure, Acute and Chronic renal failure, Nephrotic syndrome.

    * Hyperglycemia: blood glucose > 180 mg/ dl.
    * Require ICU admission.
    * Severe Protein Energy Malnutrition: Defined as grade III (50-59% of expected weight for age) and grade IV (less than 50% of expected weight for age) as per IAP classification.
    * Patients in whom either hypotonic or isotonic solutions may be contraindicated/necessary: i.e. specific neurosurgical patients (ie those at risk of increased ICP, e.g. requiring actual brain surgery, ICP monitor or external ventricular drain insertion), patients with diabetic ketoacidosis, acute (≤ 7 days) burns, pre-existing CHF, liver failure or cirrhosis, renal failure.
    * Patients with known pre-existing risk of PNa derangements: DI or SIADH

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2010-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Dicembrino, md, Principal Investigator — Hospital de Niños Pedro de Elizalde
Locations (1):
- Hospital de Niños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Choong K, Kho ME, Menon K, Bohn D. Hypotonic versus isotonic saline in hospitalised children: a systematic review. Arch Dis Child. 2006 Oct;91(10):828-35. doi: 10.1136/adc.2005.088690. Epub 2006 Jun 5. PMID 16754657
- [Background] Neville KA, Sandeman DJ, Rubinstein A, Henry GM, McGlynn M, Walker JL. Prevention of hyponatremia during maintenance intravenous fluid administration: a prospective randomized study of fluid type versus fluid rate. J Pediatr. 2010 Feb;156(2):313-9.e1-2. doi: 10.1016/j.jpeds.2009.07.059. Epub 2009 Oct 9. PMID 19818450
- [Background] Yung M, Keeley S. Randomised controlled trial of intravenous maintenance fluids. J Paediatr Child Health. 2009 Jan-Feb;45(1-2):9-14. doi: 10.1111/j.1440-1754.2007.01254.x. Epub 2007 Nov 25. PMID 18036144
- See also: Hyponatremia treatment guidelines 2007: expert panel recommendations — http://www.ncbi.nlm.nih.gov/pubmed/17981159

RESULTS

PARTICIPANT FLOW:
Groups:
- ClNa 0.3%: maintenance solution with ClNa 0.3%
- ClNa 0.45%: maintenance solution with ClNa 0.45%
Period: Overall Study
Arm/Group | ClNa 0.3% | ClNa 0.45%
Started | 42 | 36
Completed | 29 | 29
Not Completed | 13 | 7
Not completed — Protocol Violation | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ClNa 0.3% | ClNa 0.45% | Total
Number analyzed (Participants) | 42 | 36 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 36 | 78
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 105.6 (35.1) | 94.4 (42.2) | 100.5 (38.7)
Gender [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 28 | 23 | 51
Region of Enrollment [Number; unit: participants]
  Argentina | 42 | 36 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in Sodium Levels
Time Frame: Change from baseline in sodium level after 12 hours
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | ClNa 0.3% | ClNa 0.45%
Number analyzed (Participants) | 42 | 36
mEq/L
  Natremia baseline | 139.9 (3.4) | 138.1 (3.6)
  Natremia at 12 hours | 138.1 (3.4) | 138.2 (4.0)
Statistical Analysis 1: Comparison: ClNa 0.3% vs ClNa 0.45%; Serum Sodium difference at the beginning; Test type: Superiority or Other; p = 0.030, t-test, 2 sided
Statistical Analysis 2: Comparison: ClNa 0.3% vs ClNa 0.45%; Serum Sodium at the end of the study; Test type: Superiority or Other; p = 0.871, t-test, 2 sided

2. Secondary Outcome: IV Fluid Intake
Time Frame: 12 hours from baseline
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | ClNa 0.3% | ClNa 0.45%
Number analyzed (Participants) | 29 | 29
ml | 1434 (444) | 1448 (344)
Statistical Analysis 1: Comparison: ClNa 0.3% vs ClNa 0.45%; Test type: Superiority or Other; p = 0.895, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: until hospital discharge, average 5 days
Arm/Group | ClNa 0.3% | ClNa 0.45%
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 2/29 | 5/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClNa 0.3% (N=29) | ClNa 0.45% (N=29)
nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) — seizures, coma, headache.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ClNa 0.3% (N=29) | ClNa 0.45% (N=29)
hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 5 (5) — serum sodium between 130-134.9 meq/L
hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — serum sodium more than 145 mEq/L

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No